CLINICAL TRIAL: NCT03981575
Title: Establishing Biomarkers and Clinical Endpoints in Myotonic Dystrophy Type 1 (END-DM1)
Brief Title: Estab Biomarkers and Clinical Endpoints in Myotonic Dystrophy Type 1 (END-DM1)
Status: Recruiting | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: University of Rochester (Other); Stanford University (Other); Ohio State University (Other); University of Florida (Other); University of Iowa (Other); Ludwig-Maximilians - University of Munich (Other); Fondazione Serena Onlus - Centro Clinico NeMO Milano (Other); The Methodist Hospital Research Institute (Other); Radboud University Medical Center (Other); University College London Hospitals (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Other Study IDs: HM20014419; DMCRN (Other: University of Rochester); FD-R-006071 (Other Grant/Funding Number: OPD)
Record Dates: First submitted 2019-06-02; First posted 2019-06-11 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Myotonic Dystrophy 1; DM1
Keywords: Myotonic Dystrophy; END DM-1; Muscular Dystophy; DMCRN
MeSH Terms: conditions — Myotonic Dystrophy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biopsy sub-study will examine RNA splicing defects that are characteristic of DM1.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Visits: Patients will receive standard of care as determined by their treating physician. Study visits occur at baseline/0 months, 12 months, and 24 months

SUMMARY:
Building on previous work of the Myotonic Dystrophy Clinical Research Network (DMCRN), the present study seeks to overcome insufficient data on natural history; lack of reliable biomarkers; and incomplete characterization and limited biological understanding of the phenotypic heterogeneity of Myotonic Dystrophy 1 by examining strategies to improve the reliability by making further refinements in our sample collection and analysis procedures by developing strategies for managing patient heterogeneity going forward.

Funding Source- FDA OOPD

DETAILED DESCRIPTION:
Approximately 700 adult participants (18 to 70 years old, inclusive) with DM1 will be enrolled at 15 centers (up to 70 patients will be recruited at each site). No treatment will be administered as part of this study. Participants will receive standard of care as determined by the investigators. Study visits occur at baseline/0 months, 12 months, and 24 months. Few restrictions are placed on participation in the study because the investigators aim to capture the full spectrum of disease severity.

Muscle biopsy sub-study: Studies of splicing biomarkers in muscle biopsy samples will be conducted on a subset of 95 participants. These participants will have an additional study visit at 3 months.

Longitudinal muscle biopsy sub-study: Up to 30 individuals who have had a prior muscle biopsy as part of a DMCRN study will be asked to undergo another biopsy greater than 24 months after the prior biopsy. These participants will have an additional ad hoc biopsy visit.

COVID-19 sub-study: To evaluate severity of illness and response to COVID-19 vaccination in DM1 patients compared to corresponding data available about the general population, END-DM1 study participants will be asked to complete a one-time survey about COVID-19 experiences. A subset of those participants' blood samples will be analyzed to understand immunoglobulin response to infection and vaccination in DM1 patients.

Actigraphy sub-study: To assess daily physical activity in individuals with DM1 and evaluate physical activity changes over a 12-24 month period related to disease progression, a subset of participants will be asked to wear a small, wireless activity monitor while performing functional assessments described in the main study. Those participants will be asked to wear the activity monitor for 7 days following their research visit. Those participants will be asked to complete additional questionnaires.

Handheld Dynamometry sub-study: To evaluate additional muscle strength methods, a subset of participants will be asked to complete additional strength testing using either the MEDup or MicroFET handheld dynamometry device on the same day as their END-DM1 main study visit. Those participants will be asked to return to the clinic for a second visit within 10 days of the END-DM1 study visit to repeat the handheld dynamometry assessments and complete additional strength measures.

ELIGIBILITY:
Inclusion criteria:

* Age 18 to 70 (inclusive)
* Competent to provide informed consent
* Clinical diagnosis of DM1 based on research criteria1 or positive genetic test
* Comment: The clinical research criteria require myotonia, muscle weakness in a characteristic distribution, and history of similar findings in a first degree relative. Genetic testing confirmed the diagnosis of DM1 in > 99% of individuals who satisfied these criteria.2

Exclusion criteria:

* Symptomatic renal or liver disease, uncontrolled diabetes or thyroid disorder, or active malignancy other than skin cancer.
* Current alcohol or substance abuse
* Concurrent enrollment in clinical trial for DM1, or participation in trial within 6 months of entry.
* Concurrent pregnancy or planned pregnancy during the course of the study.
* Concurrent medical condition that would, in the opinion of the investigator or clinical evaluator, compromise performance on study measures.
* Note: non-ambulatory participants are not excluded, but are limited to <15% of enrollment.

Inclusion criteria for participants in the muscle biopsy sub-study:

• Of the 95 patients undergoing the tibialis anterior muscle biopsy, at least half will have at least moderate weakness of ankle dorsiflexion, defined as MRC score ≤ 4+. This is in order to obtain a muscle tissue sample in a person more severely affected with myotonic dystrophy. Approximately 10 patients at each site will undergo the muscle biopsy.

Exclusion criteria for 95 participants in the muscle biopsy sub-study:

* Known CTG repeat expansion size less than 100 repeats, unless there are clear cut signs of limb weakness and muscle wasting. This is in order to obtain a muscle tissue sample in a person more severely affected with myotonic dystrophy.
* Use of anticoagulant such as warfarin or a direct oral anticoagulant (e.g. dabigatran) due to the increased risk of bleeding.
* Use of aspirin or non-steroidal anti-inflammatory agents should be discontinued 3 days prior to the biopsy procedure, if possible.
* Platelet count <50,000 (if known) due to the increased risk of bleeding.
* History of a bleeding disorder due to the increased risk of bleeding.
* Advanced wasting of tibialis anterior (TA) muscle that precludes needle muscle biopsy in order to ensure that a sample taken would be of muscle and not just fat and fascia.
* Previous muscle biopsy of either TA in order to provide muscle tissue samples of non-biopsied muscles.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: DM1 has a prevalence rate of approximately 1 per 2,300. There are no expected gender differences. Both men and women will be selected for this study.
  Children with DM1 are not included in this project because the pathophysiological basis of congenital and childhood DM1 appears to be mechanistically distinct.
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in ambulation over 24 months as measured by the 10 meter walk (m/s). | 12 and 24 months
  10 meter walk will be measured (m/s)
Change in respiratory function over 24 months as measured by spirometry, specifically the supine forced vital capacity (FVC). | 12 and 24 months
  Supine forced vital capacity (% predicted)
Percent splicing of DM1-affected splice events | 3 months
  RNA sequenced of muscle biopsy samples collected at two different times will be combined and used to calculate a percent splicing index (PMI)

OTHER OUTCOMES:
Longitudinal Muscle Biopsy Sub-study: Characterization of RNA splicing measures over a prolonged period of time (>24 months) | 24 months
  RNA sequenced of muscle biopsy samples collected at two different times will be combined and used to calculate a percent splicing index (PMI)
Longitudinal Muscle Biopsy Sub-study: Characterization of functional endpoints over a prolonged period of time (>24 months) | 24 months
  10-meter walk/run, grip strength, ADF (ankle dorsiflexion) strength, supine FVC (forced vital capacity)
COVID-19 Sub-study: Data from DM1 patients or caregivers about COVID-19 illness and vaccination experience, severity of illness and response to vaccination in DM1 patients compared to corresponding data available about the general population. | 24 months
  To evaluate the severity and rate of COVID-19 infection in patients with DM1 compared to the general population symptomatic response to COVID-19 vaccination in DM1 patients
COVID-19 Sub-study: Immunoglobulin profile and measles titers, and COVID-19 IgG titers | 24 months
  To understand immunoglobulin response to infection and vaccination in DM1 patients
Actigraphy Sub-study: Feasibility of measuring daily physical activity in individuals with DM1 in a multi-site study | 24 months
  Participants will be asked to wear an activity monitor for 7 days following their in-clinic END-DM1 study visit to evaluate whether this type of activity monitoring is feasible in future trials.
Actigraphy Sub-study: Objective daily physical activity using wireless accelerometry (ActiGraph), and comparison to normative values and patient reported physical activity. | 24 months
  Participants will be asked to wear an activity monitor for 7 days following their in-clinic END-DM1 study visit and report physical activity, to establish physical activity data in the DM1 population.
Actigraphy Sub-study: Physical activity changes over a 12-24 month period related to disease progression. | 24 months
  Participants will wear the wireless activity monitor during the functional and strength measures, and complete additional study questionnaires at their regular END-DM1 study visits.
Handheld Dynamometry Sub-study: Inter-rater reliability, standard error of measurement, and minimal detectable change of Maximal Isometric Muscle Strength force values obtained with the MEDup and MicroFET handheld dynamometers in adults with DM1 | 24 months
  Participants will be assessed using either the MEDup or MicroFET handheld dynamometer on the same day as an END-DM1 main study visit. Participants will complete a second visit +/- 10 days from that visit where HHD will be assessed using the same HHD method (either MEDup or MicroFET) used at the HHD visit. Additional functional and strength assessments will be captured at this visit.
Handheld Dynamometry Sub-study: Comparison of quantitative muscle strength testing feasibility and validity between MEDup and MicroFET with the existing Fixed-QMT currently used in the END-DM1 study protocol. | 24 months
  Data captured for MEDup and MicroFET will be compared to data collected using the Fixed-QMT measures in the main END-DM1 study.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Johnson, MD, Principal Investigator — Virginia Commonwealth University; Charles Thornton, MD, Principal Investigator — University of Rochester
Locations (17):
- United States (10):
  - University of California, San Diego, La Jolla, California
  - University of California, Los Angeles, Los Angeles, California
  - University of Colorado - Denver, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Kansas University Medical Center, Kansas City, Kansas
  - University of Rochester, Rochester, New York
  - Ohio State University, Columbus, Ohio
  - Houston Methodist Neurological Institute, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Université de Sherbrooke, Québec, Canada
- Friedrich Baur Institute, Ludwig-Maximilians-Universität München, München, Germany
- Centro Clinico NeMO, Milan, Italy
- Radboud University Medical Center, Nijmegen, Netherlands
- University of Auckland, Auckland, New Zealand
- United Kingdom (2):
  - St. George's, University of London, London
  - University College London, London

IPD SHARING:
Plan to Share IPD: No
Aggregated and deidentified data will be shared with qualified investigators upon majority approval of the DMCRN investigators.

REFERENCES:
- [Derived] Mul K, Eichinger K, Hung M, Sansone VA, Gagnon C, Subramony S, Roxburgh RH, Hamel J, Statland JM, Elsheikh B, Turner C, Sampson J, Ragole T, Matthews E, Schoser B, Swenson A, Laverty C, Shieh P, Greene EP, Takahashi M, Wicklund M, Dekdebrun J, Raymond J, DeSpain E, Thornton CA, Johnson NE; Myotonic Dystrophy Clinical Research Network. Establishing biomarkers and clinical endpoints in myotonic dystrophy type 1 (END-DM1): Protocol of an international natural history study. PLoS One. 2025 Dec 11;20(12):e0331163. doi: 10.1371/journal.pone.0331163. eCollection 2025. PMID 41379803
- [Derived] Provenzano M, Ikegami K, Bates K, Gaynor A, Hartman JM, Jones A, Butler A, Berggren KN, Dekdebrun J, Hung M, Lapato DM, Kiefer M, Thornton CA, Johnson NE, Hale MA; Myotonic Dystrophy Clinical Research Network (DMCRN). The Splice Index as a prognostic biomarker of strength and function in myotonic dystrophy type 1. J Clin Invest. 2025 Jan 7;135(4):e185426. doi: 10.1172/JCI185426. PMID 39836447